CLINICAL TRIAL: NCT04027101
Title: BAriCitinib Healing Effect in earLy pOlymyalgia Rheumatica (BACHELOR Study)
Brief Title: BAriCitinib Healing Effect in earLy pOlymyalgia Rheumatica
Acronym: BACHELOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BACHELOR (29BRC18.0144)
Record Dates: First submitted 2019-05-16; First posted 2019-07-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Polymyalgia Rheumatic (PMR)
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: This is a multicenter double blinded randomized placebo controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral baricitinib 4mg/day for 12 weeks. Then, at week 12, if PMR-AS≤10, patients will receive baricitinib 2 mg for 12 weeks. If PMR-AS ≤10, the patients will not receive any treatment until W24 At W24, if PMR-AS>10, they will receive GCs according to the PMR-AS (PMR-AS<10: no GCs, PMR-AS between 10-20: 10mg/day, PMR-AS between 21-30: GCs at 15mg/d and if PMR-AS> 30: 20mg/d or more according to investigator's opinion). Dosage of GCs will be decreased (1 mg every week) or increased according to PMR-AS (PMR-AS < 10: decrease, PMR-AS > 20 increase, 10 ≤ PMR-AS ≤ 20: stable dose) according to investigator's opinion.
  Interventions: Drug: Baricitinib
- Control group (Placebo Comparator): Oral placebo every day during 3 months (W12). Then, at week 12, if PMR-AS ≤10, placebo for 12 weeks. If PMR-AS ≤10, the patients do not receive any treatment until a flare. If PMR-AS>10, they will receive GCs according to the PMR-AS (PMR-AS<10: no GCs, PMR-AS between 10-20: 10mg/day, PMR-AS between 21-30: GCs at 15mg/d and if PMR-AS> 30: 20mg/d or more according to investigator's opinion). Dosage of GCs will be decreased (1mg every week) or increased according to PMR-AS (PMR-AS < 10: decrease, PMR-AS > 20 increase, 10 ≤ PMR-AS ≤ 20: stable dose) and according to investigator's opinion.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Baricitinib — patient will take a tablet of 4 mg/d during 12 weeks and then 2 mg/d during 12 weeks if the patient achieves PMR-AS≤ 10 at week 12
  Arms: Experimental group
Drug: Placebos — patient will take a tablet of 4 mg/d during 12 weeks and then 2 mg/d during 12 weeks if the patient achieves PMR-AS≤ 10 at week 12
  Arms: Control group

SUMMARY:
Patients with recent PMR(6 months or less) with a PMR-AS >17 and no oral or parenteral GCs during the past 2 weeks (at least) will be included.

Treatment with oral baricitinib 4mg or placebo during 12 weeks and then, if PMR-AS≤10, they will receive baricitinib 2 mg for 12 weeks and then will stop treatment.

No rescue is allowed before week 4 (visit 3) but patients may receive up to 2 intra-articular or soft tissue injections of GCs until week 4 according to investigator's opinion.

From week 4 to week 12, steroids will be proposed as a rescue for both arms at investigators' discretion and according to PMR-AS.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age
* Fulfilling ACR/EULAR criteria for PMR
* Disease duration ≤6 months
* No oral or parenteral steroid since ≥ 2 weeks prior to randomization
* PMR-AS >17
* Absence of connective tissue diseases or vasculitis
* Able to give informed consent

Exclusion Criteria:

* Clinical symptoms of giant cell arteritis
* Uncontrolled high blood pressure or cardiovascular disease
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to PMR
* Planned major surgical procedure during the study.
* History of malignant neoplasm within the last 5 years (or 3 years in case of cervical carcinoma, basal cell or squamous epithelial skin cancer resected with no evidence of recurrence or metastatic disease).
* Current active uncontrolled infection
* Detailed exclusion criteria related to prior or concomitant therapy, general safety and laboratory data are reported in the protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Following of the Polymyalgia Rheumatica Activity score | 12 weeks
  The activity of Polymyalgia Rheumatica is evaluated using the Polymyalgia Rheumatica Activity score (PMR-AS), a disease activity score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment , Visual Analog Score for patient's pain (VAS), and CRP level. The PMR-AS is considered as relevant to define relapse and remission but also to decide if treatment have to be decreased, unchanged or increased (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose)

SECONDARY OUTCOMES:
Following of the Polymyalgia Rheumatica Activity score | 36 weeks
  The activity of Polymyalgia Rheumatica is evaluated using the Polymyalgia Rheumatica Activity score (PMR-AS), a disease activity score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment , Visual Analog Score for patient's pain (VAS), and CRP level. The PMR-AS is considered as relevant to define relapse and remission but also to decide if treatment have to be decreased, unchanged or increased (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose)
Emergence of adverse events (Safety and tolerability) | 36 weeks
  The safety is evaluated with the adverse events in both arms
Following of the cumulative dosages of Glucocorticoids | 36 weeks
  dosages of GCs
ultrasound of synovitis and tenosynovitis | 24 weeks
  ultrasound scoring of synovitis and tenosynovitis
Level of biological markers | 24 weeks
  Level of biological markers and cell subpopulations (Interleukin, cytokines, immune cells) by result of blood test is evaluated.
Following of the quality of life | 36 weeks
  The Short Form 36 (SF36) is used to evaluate the quality of life. The SF36 scale includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue].
Following of the quality of life | 36 weeks
  The Hospital Anxiety and the Depression scale (HAD) is used to evaluate the quality of life.
  The HAD scale has 14 items rated from 0 to 3 with 7 questions relate to anxiety and 7 others to the depressive dimension.
Following of the quality of life | 36 weeks
  The scale EuroQol 5 dimensions (EDQ5) is used to evaluate the quality of life. The EQ-5D scale is a standardised measure of health status to provide a simple, generic measure of health for clinical and economic appraisal, whih is divided by the EQ-5D descriptive system (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the EQ Visual Analogue scale (EQ VAS). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems).

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Chu Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CH Le Mans, Le Mans
  - CHU Montpellier, Montpellier
  - Ch Morlaix, Morlaix
  - CHU Nice, Nice
  - CHU Strasbourg, Strasbourg
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Saraux A, Carvajal Alegria G, Dernis E, Roux C, Richez C, Tison A, Quere B, Jousse-Joulin S, Guellec D, Marhadour T, Kervarrec P, Cornec D, Le Henaff C, Lesven S, Nowak E, Souki A, Devauchelle-Pensec V. Baricitinib in early polymyalgia rheumatica (BACHELOR): a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet Rheumatol. 2025 Apr;7(4):e233-e242. doi: 10.1016/S2665-9913(24)00270-4. Epub 2025 Jan 13. PMID 39818228